CLINICAL TRIAL: NCT07383870
Title: A Single-Center, Randomized, Crossover, Prospective, Open-Label, Non-Inferiority Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of an AI- and Ultrasound-Based Medical Device That Assists Venipuncture, Compared With Manual Venipuncture
Brief Title: Clinical Evaluation of an AI- and Ultrasound-Assisted Venipuncture Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: AIRS Medical Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AM-AIIV-2501; 2511-143-1698 (Other: IRB of Seoul National University Hospital)
Record Dates: First submitted 2026-01-12; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Venipuncture
Keywords: Venipuncture; Ultrasound; Artificial Intelligence; Medical device; Vascular access; Phlebotomy

STUDY DESIGN:
Intervention Model Description: This clinical trial is designed as a within-subject, randomized, crossover comparative study, in which the unit of comparison is not the subject but both arms (venipuncture sites) of each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (device-assisted venipuncture) Arm (Active Comparator): Participants will undergo venipuncture assisted by the AI- and ultrasound-based medical device (AIIV L2).
  Interventions: Device: AIIV L2
- Control (manual venipuncture) Arm (Active Comparator): Participants will undergo venipuncture using the standard manual venipuncture technique.
  Interventions: Procedure: Manual venipuncture

INTERVENTIONS:
Device: AIIV L2 — The investigational device is AIIV L2 (product code: H2BXXA2), an AI- and ultrasound-based medical device designed to assist venipuncture. This medical device is intended for use by healthcare professionals in medical institutions to obtain ultrasound images of the antecubital area of adult subjects, utilize an artificial intelligence model to identify the location of veins, and determine the insertion site of the needle to assist with venipuncture.
  Arms: Test (device-assisted venipuncture) Arm
Procedure: Manual venipuncture — Venipuncture will be performed manually according to standard clinical practice, without use of the investigational device.
  Arms: Control (manual venipuncture) Arm

SUMMARY:
Purpose

: This study aims to confirm the safety and efficacy of AIIV L2, an artificial intelligence- and ultrasound-based medical device that assists venipuncture, by comparing venipuncture performed using AIIV L2 with manual venipuncture.

Study Design : This is a single-center, randomized, crossover, prospective, open-label, non-inferiority confirmatory clinical trial.

Methods

: Each participant will undergo venipuncture on both arms: one arm using AIIV L2 and the other arm using manual venipuncture, according to randomized allocation. After venipuncture is performed on both arms, outcomes including venipuncture success rate, procedure time, pain, and hemolysis will be evaluated. All venipuncture procedures will be performed by the same operator. Vital signs and adverse events will be monitored before and after the procedure.

- Primary Efficacy Endpoint

Venipuncture success rate:

Comparison of the success rate of venipuncture on the first attempt between AI-assisted venipuncture and manual venipuncture.

- Secondary Efficacy Endpoints

Procedure time:

Time from needle insertion to completion of venipuncture.

Hemolysis rate:

Presence of hemolysis in collected samples, determined according to laboratory criteria.

Pain score (NRS):

Numeric Rating Scale (0-10) reported by participants after each venipuncture method.

Within-subject pain comparison:

Comparison of pain scores between AI-assisted and manual venipuncture within the same participant.

Acceptability:

Participant satisfaction and preference regarding AI-assisted venipuncture, assessed using a structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 19 years or older at the time of study enrollment.
* Subjects who are able to undergo venipuncture in the antecubital area of both arms, without restriction of elbow joint movement, and who can maintain the arm in a stable extended position during venipuncture.
* Subjects who have received a full explanation of the clinical trial, fully understand the contents, voluntarily decide to participate, and provide written informed consent prior to screening procedures.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Subjects with an implanted defibrillator or pacemaker.
* Subjects at increased risk of bleeding due to underlying conditions such as anticoagulant use, hemophilia, thrombocytopenia, preeclampsia, or other coagulation disorders.
* Subjects with abnormal vascular anatomy in the antecubital area due to vascular malformations, vascular disease, or prior creation of an arteriovenous shunt.
* Subjects with significant abnormal skin lesions (e.g., infection, dermatologic disease, trauma, or wounds) in the antecubital area.
* Subjects whose arm condition is unsuitable for venipuncture due to transfusion, intravenous fluid therapy, or similar procedures.
* Subjects with immunodeficiency or immunosuppression (e.g., steroid or immunosuppressant therapy, severe infection) and therefore vulnerable to infection.
* Subjects with a prior history of severe vasovagal reaction during venipuncture.
* Subjects whose upper arm circumference exceeds 44 cm, preventing application of the tourniquet inside the device.
* Subjects with a conflict of interest, such as employees of competing companies.
* Subjects considered by the investigator to be otherwise unsuitable for participation in this clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
First-attempt venipuncture success rate | Immediately after venipuncture
  First-attempt venipuncture success is defined as successful collection of at least 1 mL of blood into a collection tube at the first needle insertion into the participant's arm.

SECONDARY OUTCOMES:
Procedure time | During each venipuncture procedure
  Procedure time is defined as the duration that directly affects the participant. The measurement start time is defined as the moment of first direct contact with the participant after completion of subject verification and preparation of consumables.
  For device-assisted venipuncture, the start time is defined as the time point at which the "search start" button is pressed and the tourniquet is automatically applied. For manual venipuncture, the start time is defined as the earlier of the time point when the tourniquet is applied by the operator or when the operator begins palpation of the vein.
  For both methods, the measurement end time is defined as the time point at which venipuncture is completed and hemostasis is initiated.
Hemolysis Rate | Assessed by analyzing the blood samples obtained after venipuncture.
  Hemolysis is objectively assessed for all collected blood samples using an automated hemolysis index. Hemolysis is defined as a hemoglobin concentration greater than 0.5 g/L.
Pain score during device-assisted venipuncture (NRS) | Immediately after device-assisted venipuncture
  Pain intensity experienced by participants during device-assisted venipuncture is assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain).
Comparative pain assessment versus manual venipuncture | Immediately after completion of both venipuncture procedures
  Participants subjectively compare pain experienced during device-assisted venipuncture relative to manual venipuncture, categorized as "less painful," "similar," or "more painful."
Acceptability of device-assisted venipuncture | Immediately after completion of both venipuncture procedures
  Acceptability of device-assisted venipuncture is assessed by asking participants whether they would be willing to undergo venipuncture using the device again in the future.
Incidence of venipuncture-related adverse events | Immediately after venipuncture and during the short-term observation period
  Incidence of adverse events related to venipuncture assessed immediately after the procedure and during the short-term observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Song, MD, PhD, Principal Investigator — Seoul National University Hospital / Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No